CLINICAL TRIAL: NCT02763969
Title: Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986202 in Healthy Subjects and to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Efficacy of BMS-986202 in Subjects With Moderate to Severe Psoriasis
Brief Title: Safety Study of BMS-986202 in Healthy Subjects and to Treat Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM016-006
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — BMS-986202; Interferon alpha-2; Famotidine; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A: Single Ascending Dose (Experimental): BMS-986202 or Placebo specified dose on specified days
  Interventions: Drug: BMS-986202; Drug: Placebo
- Part B: Multiple Ascending Dose (Experimental): BMS-986202 or Placebo + Interferon alpha-2a recombinant specified dose on specified days
  Interventions: Drug: BMS-986202; Drug: Placebo; Drug: Interferon alpha-2a recombinant
- Part C: Multiple Ascending Dose-Japanese descent (Experimental): BMS-986202 or Placebo specified dose on specified days in patients of Japanese descent
  Interventions: Drug: BMS-986202; Drug: Placebo
- Part D: Relative Bioavailability (Experimental): BMS-986202 (Liquid) or BMS-986202 (Capsule) + Famotidine specified dose on specified days
  Interventions: Drug: BMS-986202; Drug: Famotidine
- Part E: Proof of Mechanism (Experimental): BMS-986202 or Placebo + Ustekinumab specified dose on specified days
  Interventions: Drug: BMS-986202; Drug: Placebo; Drug: Ustekinumab

INTERVENTIONS:
Drug: BMS-986202
Drug: Placebo
  Arms: Part A: Single Ascending Dose; Part B: Multiple Ascending Dose; Part C: Multiple Ascending Dose-Japanese descent; Part E: Proof of Mechanism
Drug: Interferon alpha-2a recombinant
  Arms: Part B: Multiple Ascending Dose
Drug: Famotidine
  Arms: Part D: Relative Bioavailability
Drug: Ustekinumab
  Arms: Part E: Proof of Mechanism

SUMMARY:
The purpose of this study is to establish if BMS-986202 is safe and effective at treating autoimmune diseases such as psoriasis. BMS-986202 which has shown some promise in preclinical studies for inhibiting autoimmune conditions such as psoriasis. This study will be the first time this drug is given to humans.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy Male and Female participants
* 18 to 50 years of age (Parts A-D)
* 18 to 70 years of age (Part E)
* Diagnosed with plaque psoriasis (Part E)

Exclusion Criteria:

* Participants that had recent infections
* Participants with Low Blood Pressure
* Participants with any heart related problems
* Participants with cancer
* Participants with any other major medical illness

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Safety of a single oral dose of BMS-986202 based on number of incidence of AEs, SAEs, AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | 4 weeks after the start of treatment
Safety of a multiple oral dose of BMS-986202 based on number of incidence of AE, SAEs, AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations | 4 weeks after the start of treatment
Change from baseline in the psoriasis area | 4 weeks after the start of treatment
Severity index (PASI) score | 4 weeks after the start of treatment

SECONDARY OUTCOMES:
Effect of BMS-986202 on electrocardiographic (ECG) parameters such as heart rate in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
Effect of BMS-986202 on electrocardiographic (ECG) parameters such as PR interval in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
  The interval from the beginning of the P wave to the beginning of the QRS complex (PR interval)
Effect of BMS-986202 on electrocardiographic (ECG) parameters such as QRS interval in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
  The interval from the beginning of the Q wave and the end of the S wave (QRS interval)
Effect of BMS-986202 on electrocardiographic (ECG) parameters such as QTc interval in healthy subjects of any ethnic background (Parts A, B, C, D) | Approximately 3 months
  The interval from the beginning of the Q wave to the end of the T wave (QT interval).
  The QT interval corrected for heart rate (QTc interval)
Safety of multiple oral doses of BMS-986202 in subjects with moderate to severe psoriasis (Part E) | Approximately 3 months
  Safety of multiple oral doses of BMS-986202 in subjects with moderate to severe psoriasis (Part E) based on number of incidence of adverse events(AEs), serious adverse events(SAEs), AEs leading to discontinuation or death, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, telemetry, and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Australia (2):
  - Local Institution, Melbourne, Victoria
  - Local Institution, Melbourne

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx